CLINICAL TRIAL: NCT04882423
Title: Effect of Vegetable Intake on Heterocyclic Amine Metabolism in Humans
Brief Title: Vegetable Intake Effect on Heterocyclic Amine Metabolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the university
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2013NTLS067
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer
Keywords: HAA; Heterocyclic aromatic amines; apiaceous vegetables; cruciferous vegetables
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: In a randomized crossover design, each participant will undergo four study phases with a different test meal at the end of each phase. Every phase will consist of subjects consuming for six days their normal diet excluding cruciferous and apiaceous vegetables, alcohol, and caffeine. Furthermore, participants will refrain from meat products for 24 hours prior to the test meal, given that HAA are generally excreted in the urine by 12 hours post ingestion (18, 80). Compliance will be assessed with a questionnaire and the analysis of baseline levels of phytochemicals in spot urine samples that are to be collected prior to the test meal. On day seven of each phase and after an overnight fast, subjects will be randomly assigned to eat (in a private room near Dr. Truda's lab) one of four meals (prepared in a food grade lab also near Dr. Truda's lab)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test meal 1 - grilled hamburger (7 oz) with no vegetables (Experimental): Randomly assigned participants are given grilled hamburger (7 oz) with no vegetables
  Interventions: Other: grilled hamburger (7 oz) with no vegetables
- Test meal 2 - grilled hamburger with steamed broccoli and Brussels sprouts (Experimental): Randomly assigned participants are given grilled hamburger with steamed broccoli and Brussels sprouts (3g/kg body weight combined)
  Interventions: Other: grilled hamburger (7 oz) with steamed broccoli and Brussels sprouts (3g/kg body weight combined)
- Test meal 3 - grilled hamburger with steamed parsnips, fresh parsley, and celery sticks (Experimental): Randomly assigned participants are given grilled hamburger (7 oz) with steamed parsnips, fresh parsley, and celery sticks (3g/kg body weight combined)
  Interventions: Other: grilled hamburger (7 oz) with steamed parsnips, fresh parsley, and celery sticks (3g/kg body weight combined)
- Test meal 4- grilled hamburger with broccoli, Brussels sprouts, parsnips, parsley and celery sticks (Experimental): Randomly assigned participants are given grilled hamburger (7 oz) with steamed broccoli, Brussels sprouts, and parsnips plus fresh parsley and celery sticks (6g/kg body weight combined).
  Interventions: Other: grilled hamburger (7 oz) with steamed broccoli, Brussels sprouts, and parsnips plus fresh parsley and celery sticks (6g/kg body weight combined).

INTERVENTIONS:
Other: grilled hamburger (7 oz) with no vegetables — Test meal 1: grilled hamburger (7 oz) with no vegetables
  Arms: Test meal 1 - grilled hamburger (7 oz) with no vegetables
Other: grilled hamburger (7 oz) with steamed broccoli and Brussels sprouts (3g/kg body weight combined) — Test meal 2: grilled hamburger (7 oz) with steamed broccoli and Brussels sprouts (3g/kg body weight combined)
  Arms: Test meal 2 - grilled hamburger with steamed broccoli and Brussels sprouts
Other: grilled hamburger (7 oz) with steamed parsnips, fresh parsley, and celery sticks (3g/kg body weight combined) — Test meal 3: grilled hamburger (7 oz) with steamed parsnips, fresh parsley, and celery sticks (3g/kg body weight combined)
  Arms: Test meal 3 - grilled hamburger with steamed parsnips, fresh parsley, and celery sticks
Other: grilled hamburger (7 oz) with steamed broccoli, Brussels sprouts, and parsnips plus fresh parsley and celery sticks (6g/kg body weight combined). — Test meal 4: grilled hamburger (7 oz) with steamed broccoli, Brussels sprouts, and parsnips plus fresh parsley and celery sticks (6g/kg body weight combined).
  Arms: Test meal 4- grilled hamburger with broccoli, Brussels sprouts, parsnips, parsley and celery sticks

SUMMARY:
This is a randomized trial with crossover design, where each participant will undergo four study phases with a different test meal at the end of each phase. Every phase will consist of subjects consuming for six days their normal diet excluding cruciferous and apiaceous vegetables, alcohol, and caffeine. The participants will refrain from meat products for 24 hours prior to the test meal. On day seven of each phase and after an overnight fast, subjects will be randomly assigned to eat one of four meals:

1. grilled hamburger with no vegetables
2. grilled hamburger with steamed broccoli and Brussels sprouts
3. grilled hamburger with steamed parsnips, fresh parsley, and celery sticks
4. grilled hamburger with steamed broccoli, Brussels sprouts, and parsnips plus fresh parsley and celery sticks.

DETAILED DESCRIPTION:
Colon cancer is the third most common cancer in the U.S. Convincing evidence suggests that high intake of red meat increases colon cancer risk, according to the 2007 AICR/WCRF Second Expert Report. The likely responsible mutagens are heterocyclic aromatic amines (HAA), which form naturally during the cooking of meat, poultry, and fish at high temperatures. Bioactivation of HAA to carcinogenic metabolites is primarily mediated by phase I biotransformation enzymes. Evidence suggests that the activity of many of these enzymes can be modulated by constituents in apiaceous vegetables (parsnips, celery, etc.) and cruciferous vegetables (broccoli, cabbage, etc.)

In this trial researchers are comparing the effects of eating cruciferous vegetables, apiaceous vegetables, or both groups combined on HAA metabolism after eating grilled hamburger together in a single meal. They aim to define optimal dietary patterns and food combinations that maximize the safe excretion of dietary carcinogens through this trial. This contribution is significant because the knowledge gained will be applicable to the prevention of colon cancer as well as additional cancers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Healthy
* Non-smoker

Exclusion Criteria:

* No history of gastrointestinal, hepatic, or renal disorders
* Not currently taking any prescription or over-the-counter medications
* Not currently taking any herbal/vitamins supplements
* Not pregnant or lactating
* No allergies or intolerances to the foods that will be used in the study (parsnips, parsley, celery, broccoli, Brussels sprouts, and hamburger)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Hydroxylated PhlP profile with cruciferous vegetables | 24 hours
  Quantify Hydroxylated PhlP in ng per ml of urine will be measured using LC-MS metabolomics approach.
Hydroxylated PhlP profile with apiaceous vegetables | 24 hours
  Quantify Hydroxylated PhlP in ng per ml of urine will be measured using LC-MS metabolomics approach.
Hydroxylated PhlP profile with both cruciferous and apiaceous vegetables | 24 hours
  Quantify Hydroxylated PhlP in ng per ml of urine will be measured using LC-MS metabolomics approach.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Trudo, PhD, RD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States